CLINICAL TRIAL: NCT03363581
Title: Food Preference Following Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Carel Le Roux, Reader in Investigative Science, Imperial College London
Other Study IDs: GutHormoneStudy
Record Dates: First submitted 2017-08-09; First posted 2017-12-06 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2022-10

CONDITIONS: Obesity
Keywords: Food preferences; Fat; Weight loss
MeSH Terms: conditions — Obesity; Food Preferences; Platelet Glycoprotein IV Deficiency; Weight Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood- Plasma and Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric bypass: Obese patients due to undergo gastric bypass surgery
  Interventions: Behavioral: Food Preference
- Control: Healthy free-living individuals
  Interventions: Behavioral: Food Preference

INTERVENTIONS:
Behavioral: Food Preference — Buffet meal to assess food preference

SUMMARY:
Roux-en-Y gastric bypass (RYGB) decreases appetite, caloric intake, glycemia, and body weight, all of which are maintained long term.It is controversial whether, after RYGB, patients choose to eat less high fat and sugary foods in favor of lower energy dense alternatives. Therefore the proposition to use direct measures in humans after RYGB to test the hypothesis that the selection and intake of foods varying in fat content and glycemic index, as well as the pattern of ingestion within and across meals, changes in a manner that leads to beneficial outcomes on body weight.

DETAILED DESCRIPTION:
Roux-en-Y gastric bypass (RYGB) decreases appetite, caloric intake, glycemia, and body weight, all of which are maintained long term.It is controversial whether, after RYGB, patients choose to eat less high fat and sugary foods in favor of lower energy dense alternatives. If true, this could conceivably contribute to improved glycemia and body weight. Disparities among studies on food selection and intake are likely due to the almost complete reliance on self-reported food intake which is vulnerable to inaccuracy.This controversy can best be resolved by complementing existing findings with direct measures of target behaviour in humans. Therefore the proposition to use direct measures in humans after RYGB to test the hypothesis that the selection and intake of foods varying in fat content and glycemic index, as well as the pattern of ingestion within and across meals, changes in a manner that leads to beneficial outcomes on body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Surgical and non-surgical groups:

   A) Bariatric surgery B) Controls with no history of bariatric surgery
2. Independently mobile
3. Capacity to consent to participate
4. >18 years of age

Exclusion Criteria:

1. Pre-operatively: significant dysphagia, gastric outlet obstruction or anything that prevents subjects from eating a meal.
2. Post-operatively: significant and persistent surgical complications or anything that prevents subjects from eating a meal.
3. Systemic or gastrointestinal condition which may affect food intake or preference, including:

   i) pregnancy or ii) breast feeding.
4. Active and significant psychiatric illness including substance misuse
5. Significant cognitive or communication issues
6. Medications with documented effect on food intake or food preference
7. History of significant food allergy and certain dietary restrictions
8. History of liver disease or pancreatitis
9. History of bradyarrythmia or congestive cardiac failure group)
10. Use of medications with potential serious interactions with Octreotide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with obesity attending a specialist obesity clinic and free living individuals.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carel le Roux, MBChB, PhD, Principal Investigator — Imperial College London
Locations (1):
- University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Gastric Bypass: Patients with obesity due to undergo gastric bypass surgery
  Food Preference: Buffet meal to assess food preference
- Healthy Free-living Individuals: Healthy free-living individuals
  Food Preference: Buffet meal to assess food preference
Period: Overall Study
Arm/Group | Gastric Bypass | Healthy Free-living Individuals
Started | 14 | 20
Completed | 14 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gastric Bypass | Healthy Free-living Individuals | Total
Number analyzed (Participants) | 14 | 20 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (7.8) | 28 (4.1) | 39.5 (5.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 4 | 8 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 20 | 34
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Ireland | 14 | 20 | 34
Body weight (kg) [Mean (Standard Deviation); unit: kg] | 136 (23.8) | 65 (5.2) | 100.5 (14.5)
Total Food Intake (Lunch Buffet) [Mean (Standard Deviation); unit: kJ] — The total Intake is calculated based on energy from Fat, Protein, and Carbs. The breakdown includes the energy consumed from Simple Sugar (part of total carbohydrates).
  kJ | 6510.3 (1023) | 800 (50) | 3655 (536.5)
Absolute intake of fat [Mean (Standard Deviation); unit: kJ] | 2617.1 (250) | 310 (30) | 1448.5 (265)
Absolute intake of carbohydrates [Mean (Standard Deviation); unit: kJ] | 3102.4 (1080) | 300 (70) | 1701.2 (575)
Absolute intake of protein [Mean (Standard Deviation); unit: kJ] | 833.9 (87.0) | 190 (15) | 511.95 (94.5)
Absolute intake of sugar [Mean (Standard Deviation); unit: kJ] | 1312.5 (300) | 180 (30) | 746.25 (315)

OUTCOME MEASURES:

1. Primary Outcome: Total Food Intake (Lunch Buffet) at 24 Months
Description: Determine the effect of RYGB on total food intake from an ad libitum lunch buffet
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: kJ
Arm/Group | Gastric Bypass | Healthy Free-living Individuals
Number analyzed (Participants) | 14 | 20
kJ | 2540.1 (431.0) | 721 (201)

2. Primary Outcome: Change in Absolute Intake of Fat
Description: Determine the effect of RYGB on food preferences by measuring the absolute i.e. total intake of fat from an ad libitum lunch buffet
Time Frame: 24 months
Measure: Mean (Standard Error); unit: kJ
Arm/Group | Gastric Bypass | Healthy Free-living Individuals
Number analyzed (Participants) | 14 | 20
kJ | -1549.7 (298.9) | 301 (70.1)

3. Primary Outcome: Change in Absolute Intake of Carbohydrates
Description: Determine the effect of RYGB on food preferences by measuring the absolute i.e. total intake of carbohydrates from an ad libitum lunch buffet
Time Frame: 24 months
Measure: Mean (Standard Error); unit: kJ
Arm/Group | Gastric Bypass | Healthy Free-living Individuals
Number analyzed (Participants) | 14 | 20
kJ | -2088.6 (370.1) | 280 (40.3)

4. Primary Outcome: Change in Absolute Intake of Sugar
Description: Determine the effect of RYGB on food preferences by measuring the absolute i.e. total intake of sugar from an ad libitum lunch buffet
Time Frame: 24 months
Measure: Mean (Standard Error); unit: kJ
Arm/Group | Gastric Bypass | Healthy Free-living Individuals
Number analyzed (Participants) | 14 | 20
kJ | -890.7 (258.1) | 160.0 (39.8)

5. Primary Outcome: Change in Absolute Intake of Protein
Description: Determine the effect of RYGB on food preferences by measuring the absolute i.e. total intake of protein from an ad libitum lunch buffet
Time Frame: 24 months
Measure: Mean (Standard Error); unit: kJ
Arm/Group | Gastric Bypass | Healthy Free-living Individuals
Number analyzed (Participants) | 14 | 20
kJ | -360.7 (91.4) | 140.2 (35.2)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Gastric Bypass | Healthy Free-living Individuals
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/20
Other Adverse Events (participants affected / at risk) | 0/14 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT03363581/Prot_SAP_000.pdf
  • Informed Consent Form (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT03363581/ICF_001.pdf